CLINICAL TRIAL: NCT03956511
Title: Integrated Prediction of Extubation Outcome by the Spontaneous Breathing Trial in Newborn Infants
Status: Completed | Type: Observational
Sponsor: Ourania Kaltsogianni (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor-Investigator, Ourania Kaltsogianni, Dr Ourania Kaltsogianni, MSc Advanced Paediatrics, King's College Hospital NHS Trust
Organization: King's College Hospital NHS Trust (Other)
Other Study IDs: 193377
Record Dates: First submitted 2016-08-30; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Infant, Newborn, Diseases; Airway Morbidity
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Spontaneous Breathing Trial — It involves placing an infant from invasive mechanical pressure limited time cycled ventilation ventilation to endotracheal continuous positive end-expiratory pressure (ET-CPAP) for a period of 5 minutes during which saturation and heart rate are closely monitored. The infant would pass the test if there is no hypoxia or bradycardia during the test. If the infant has either bradycardia for more than 15 seconds and/or a fall in SpO2 below 85% despite a 15% increase in FIO2, the study will be stopped and ventilation will be restarted.

SUMMARY:
Prolonged mechanical ventilation (MV) is associated with significant adverse effects in newborn infants and clinicians aim at its minimum possible duration. Failed extubation and need for reintubation is common and further prolongs the duration of MV. Hence, accurate prediction of readiness for extubation would incur a considerable reduction in respiratory morbidity.

The Spontaneous breathing Trial (SBT) involves placing the infant on endotracheal continuous positive airway pressure for five minutes with continuous monitoring of heart rate and oxygen saturation levels. The infant would pass the test if there is no hypoxia or bradycardia during the trial. A successful SBT might predict successful extubation.

The respiratory muscles play a crucial role in successful extubation. One simple way to quantify respiratory muscle function is the rate of relaxation of the inspiratory muscles that can be depicted by the rate of the decline of the airway pressure signal following a spontaneous breath.

The hypothesis of the investigator is that respiratory muscle function assessment using the rate of relaxation of the inspiratory muscles during a SBT can accurately predict extubation outcomes either independently or in conjunction with the outcome of the SBT and the variability of the respiratory parameters during the SBT. This could increase the predicting accuracy of extubation outcomes and thus reduce re-intubation associated respiratory morbidity.

DETAILED DESCRIPTION:
Prolonged endotracheal mechanical ventilation has significant adverse effects in newborn infants including subglottic stenosis, bacterial colonisation and bronchopulmonary dysplasia. Neonatal health professionals aim to limit the period of mechanical ventilation to the minimum possible duration. The decision to extubate is commonly a clinical one, based on current ventilator settings, blood gases analysis and the overall clinical condition of the infant. On the other hand, newborn infants commonly fail extubation and require reintubation which is a traumatic invasive procedure which could further prolong the total duration of invasive mechanical ventilation. Thus, accurate prediction of readiness for extubation outcome will probably incur a notable reduction in respiratory morbidity.

A number of studies have evaluated methods to predict extubation outcome. Of them, the spontaneous breathing trial (SBT) has been shown to hold the highest predictive value: it involves placing an infant from invasive mechanical pressure limited time cycled ventilation ventilation to endotracheal continuous positive end-expiratory pressure (ET-CPAP) for a period of 5 minutes during which saturation and heart rate are closely monitored. The infant would pass the test if there is no hypoxia or bradycardia during the test. A successful SBT has a positive predictive value of 93%, sensitivity of 97% and specificity of 73%. The combination of a successful SBT with increased variability in respiratory parameters during the SBT has been reported to further increase the sensitivity of the trial; alas the specificity remains below 75%.

It should be noted that at King's College Hospital the SBT forms part of routine clinical care as per clinical guideline and it is at the discretion of the attending physician to conduct the trial prior to extubation.

The work of breathing is undertaken by the respiratory muscles. Impaired respiratory muscle function is associated with a higher risk of respiratory muscle fatigue and respiratory failure and need for mechanical ventilation. Respiratory muscle function has been identified as an independent predictor of extubation outcome in mechanically ventilated infants. One simple way to quantify respiratory muscle function is the rate of relaxation of the inspiratory muscles which can be depicted by the rate of the decline of the airway pressure signal following a spontaneous breath. In concept, inefficient muscle function is manifested by a more gradual drop to baseline of the airway pressure over time. The principle on which the method is based is that when skeletal muscles contract against increased external loads, their relaxation slows as a result of slower calcium uptake by skeletal muscle fibres. In terms of physical properties, fatigued muscle fibres take longer to relax after contraction and this reduction in the relaxation rate can be quantified by an increase in the time constant of relaxation and a decrease in the maximal relaxation rate.

The rate of relaxation of the inspiratory muscles has been shown to accurately describe respiratory muscle function in non-neonatal populations. The information on the inspiratory muscle rate of relaxation is readily available in the ventilator graphics which, as part of routine clinical care, use a pressure port and a flow sensor to record airway flow, delivered volume and pressure over time. To the knowledge of the investigator, the potential value of this information in predicting extubation outcome in newborn infants has not been explored to date.

Typically, respiratory muscle dysfunction would occur in premature infants owing to immaturity, decreased muscle mass and prematurity-associated co-morbidities. Furthermore infants with Congenital Diaphragmatic Hernia (CDH) and Anterior Wall Defects (AWD) such as gastroschisis and exomphalos, have also been reported to have impaired respiratory muscle function which could probably preclude timely successful extubation. King's College Hospital provides care for a large number of infants with CDH and AWD while also has a long tradition in the assessment of respiratory muscle function in infants making it the ideal site to recruit infants with CDH and AWD.

The hypothesis of the investigator is that respiratory muscle function assessment using the rate of relaxation of the inspiratory muscles during SBT can accurately predict extubation outcome. This prediction might stand independently for the rate of relaxation or in conjunction with SBT-derived respiratory function parameters such as the outcome of the SBT and the variability of respiratory parameters during the SBT. An integrated algorithm incorporating respiratory muscle function data could thus be produced. This would be validated in a large cohort and could increase the prediction accuracy of extubation outcome and thus reduce re-intubation associated respiratory morbidity.

This will be a prospective, observational cohort study. Aims of the study are to measure the rate of relaxation, airway flow, airway pressure, tidal volume and transcutaneous oxygen saturation in all planned extubations over the coming 12 months in the neonatal unit at King's College Hospital. Data to be recorded include basic epidemiologic parameters such as gestation at birth, birth weight, corrected gestational age at measurement, day of life, weight at measurement, blood gas parameters within 6 hours of the SBT and associated co-morbidities that might impact on the success of the SBT such as open ductus arteriosus and current evidence of infection. Infants with known genetic or chromosomal abnormalities, infants with congenital anomalies other than CDH or AWD and infants with focal acute lung pathology such as atelectasis or pneumothorax will be excluded from the study.

Based on the unit's activity over the past two chronological years, the investigators anticipate that with a successful consent rate of 80% it will be possible to measure 100 infants in total: 40 premature infants, 40 term infants and 20 infants with CDH and AWD. As this is a novel index, direct power calculation cannot be undertaken before the commencement of the study. An interim power calculation based on pilot data will be conducted half way through the project at six months, to determine the required sample size. The investigators believe however, that given that previous studies with similar outcome measures incorporated significantly smaller numbers of participants, the achieved sample size will be sufficient for the objectives of the study to be achieved.

Inform written consent will be requested from the parents or legal guardians of the infants and the attending Neonatal Consultant will be requested to assent to the study.

When the clinical team decides an infant is ready for extubation, the investigator will switch the ventilator to ET-CPAP at the same pressure as the positive end expiratory pressure during mechanical ventilation. Airflow, integrated tidal volume and airway pressure will be recorded with the NM3 respiratory function monitor (Philips Respironics, Connecticut, USA). The monitor will be connected to a Laptop (Dell Latitude, Dell, Bracknell, UK) with customised Spectra software (3.0.1.4) (Grove Medical, London, UK). The NM3 respiratory profile monitor has a combined pressure, flow and carbon dioxide sensor and this will be placed in line between the inspiratory limb of the ventilator circuit and the endotracheal tube. The NM3 monitor is automatically calibrated for flow and pressure. Flow will be measured using a fixed orifice pneumotachograph. One of the tubes from the pneumotachograph will be connected to a second pressure transducer to measure airway pressure. Oxygen saturation and heart rate monitoring will also be performed.

A failed SBT will be recorded if the infant has either a bradycardia for more than 15 seconds and/or a fall in SpO2 below 85% despite a 15% increase in FIO2. At this point the study will be stopped and ventilation will be restarted.

Infants will be extubated to either nasal CPAP or high flow nasal cannula oxygen at the clinician's discretion.

The primary study outcome will be reintubation within 72 hours of extubation. The indications for reintubation will be: (a) more than six episodes of apnoea requiring stimulation in six hours, or more than one significant episode of apnoea requiring bag and mask ventilation; (b) respiratory acidosis: PaCO2 >8.5 kPa and pH,7.25; (c)FIO2>0.60 to maintain SpO2 in the range of 90-95%.

If the infant has either bradycardia for more than 15 seconds and/or a fall in SpO2 below 85% despite a 15% increase in FIO2, the study will be stopped and ventilation will be restarted. Strict infection control policies will be followed according to the unit's guidelines.

Data will be stored until the child is 25 years old. Continuous outcomes will be compared between premature and term infants and between term infants and infants with CDH/AWD. Student's t test will be used when the data are normally distributed and Mann-Whitney U test when skewed. Categorical data will be assessed using the Fisher two tailed exact test. P<0.05 will be considered significant. The ability of respiratory variables to accurately discriminate between successful and failed extubation will be assessed using receiver operating characteristic curves. A value of the area under the curve of 0.5 will indicate no discriminatory value, and a value >0.8 will suggest a high predictive value. Standard formulae will be used to calculate sensitivity, specificity, and positive and negative predictive values and likelihood ratios. Statistical analyses will be performed using SPSS software (SPSS Inc, Chicago, Illinois, USA).

The investigators anticipate that by incorporating information on respiratory muscle function during the SBT, it will be possible to create an algorithm that will accurately predict extubation outcome in mechanically ventilated infants. The investigators also want to demonstrate that the rate of respiratory muscle relaxation might be different in premature infants, in full-term infants and in infants with surgically corrected anomalies such as CDH and AWD. These results will be incorporated in local clinical practice and form a guideline on "when to safely extubate" infants on mechanical ventilation. This will reduce respiratory morbidity associated both with prolonged ventilation as well as with failed extubation and re-intubation.

ELIGIBILITY:
Inclusion Criteria:

* All infants with a planned extubation.

Exclusion Criteria:

* Infants with known genetic or chromosomal abnormalities.
* Infants with congenital anomalies other than Congenital Diaphragmatic Hernia or Anterior Wall Defect and
* Infants with focal acute lung pathology such as atelectasis or pneumothorax will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants with a planned extubation during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Reintubation within 72 hours from extubation | Through study completion, an average one year
  Reintubation will be assessed by reviewing infant's ventilation state
Reintubation within 72 hours from extubation | Through study completion, an average one year
  Reintubation will be assessed by reviewing infant's clinical records

SECONDARY OUTCOMES:
Comparison of the rate of relaxation of respiratory muscles between premature infants that fail extubation and premature infants that successfully wean off mechanical ventilation. | Through study completion, an average one year
  Calculation of the time constant of relaxation that is the reciprocal of the slope of the decline in pressure as a function of time during the spontaneous breathing trial.
Comparison of the rate of relaxation of respiratory muscles between premature infants and term infants. | Through study completion, an average one year
  Calculation of the time constant of relaxation that is the reciprocal of the slope of the decline in pressure as a function of time during the spontaneous breathing trial.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Dassios, Consultant, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamlin CO, Davis PG, Morley CJ. Predicting successful extubation of very low birthweight infants. Arch Dis Child Fetal Neonatal Ed. 2006 May;91(3):F180-3. doi: 10.1136/adc.2005.081083. Epub 2006 Jan 12. PMID 16410255
- [Background] Stefanescu BM, Murphy WP, Hansell BJ, Fuloria M, Morgan TM, Aschner JL. A randomized, controlled trial comparing two different continuous positive airway pressure systems for the successful extubation of extremely low birth weight infants. Pediatrics. 2003 Nov;112(5):1031-8. doi: 10.1542/peds.112.5.1031. PMID 14595042
- [Background] Currie A, Patel DS, Rafferty GF, Greenough A. Prediction of extubation outcome in infants using the tension time index. Arch Dis Child Fetal Neonatal Ed. 2011 Jul;96(4):F265-9. doi: 10.1136/adc.2010.191015. Epub 2010 Nov 20. PMID 21097837
- [Background] Dimitriou G, Fouzas S, Vervenioti A, Tzifas S, Mantagos S. Prediction of extubation outcome in preterm infants by composite extubation indices. Pediatr Crit Care Med. 2011 Nov;12(6):e242-9. doi: 10.1097/PCC.0b013e3181fe3431. PMID 21037500
- [Background] Kavvadia V, Greenough A, Dimitriou G. Prediction of extubation failure in preterm neonates. Eur J Pediatr. 2000 Apr;159(4):227-31. doi: 10.1007/s004310050059. PMID 10789923
- [Background] Mikhno A, Ennett CM. Prediction of extubation failure for neonates with respiratory distress syndrome using the MIMIC-II clinical database. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:5094-7. doi: 10.1109/EMBC.2012.6347139. PMID 23367074
- [Background] Kaczmarek J, Kamlin CO, Morley CJ, Davis PG, Sant'anna GM. Variability of respiratory parameters and extubation readiness in ventilated neonates. Arch Dis Child Fetal Neonatal Ed. 2013 Jan;98(1):F70-3. doi: 10.1136/fetalneonatal-2011-301340. Epub 2012 May 3. PMID 22556206
- [Background] Kyroussis D, Mills G, Hamnegard CH, Wragg S, Road J, Green M, Moxham J. Inspiratory muscle relaxation rate assessed from sniff nasal pressure. Thorax. 1994 Nov;49(11):1127-33. doi: 10.1136/thx.49.11.1127. PMID 7831629
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Dassios T, Kaditis A, Katelari A, Chrousos G, Doudounakis S, Dimitriou G. Time constant of inspiratory muscle relaxation in cystic fibrosis. Pediatr Res. 2015 Apr;77(4):541-5. doi: 10.1038/pr.2015.2. Epub 2015 Feb 2. PMID 25642662
- [Background] Kyroussis D, Johnson LC, Hamnegard CH, Polkey MI, Moxham J. Inspiratory muscle maximum relaxation rate measured from submaximal sniff nasal pressure in patients with severe COPD. Thorax. 2002 Mar;57(3):254-7. doi: 10.1136/thorax.57.3.254. PMID 11867831
- [Background] Kassim Z, Moxham J, Davenport M, Nicolaides K, Greenough A, Rafferty GF. Respiratory muscle strength in healthy infants and those with surgically correctable anomalies. Pediatr Pulmonol. 2015 Jan;50(1):71-8. doi: 10.1002/ppul.23007. Epub 2014 Feb 20. PMID 24574153